CLINICAL TRIAL: NCT01160913
Title: Evaluation of Optimal Anatomical Layer for Continuous Wound Infusion of Local Anesthetics Combined With NSAIDs Through a Multiorifice Catheter for Postoperative Pain Intensity After Elective Cesarean Delivery
Brief Title: Optimal Site of Administration for Continuous Wound Infusion After Cesarean Section
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Association pour la Recherche et la Formation en Anesthésie Analgésie Réanimation (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KTCESAR
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2007-09

CONDITIONS: Cesarean Section

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous wound infusion above the fascia (Active Comparator)
  Interventions: Procedure: Continuous wound infusion
- Continuous wound infusion below the fascia (Active Comparator)
  Interventions: Procedure: Continuous wound

INTERVENTIONS:
Procedure: Continuous wound infusion
  Arms: Continuous wound infusion above the fascia
Procedure: Continuous wound
  Arms: Continuous wound infusion below the fascia

SUMMARY:
The purpose of this randomized double-blind study is to evaluate in which anatomical layer (AF versus BF) continuous wound infusion of local anesthetics combined with NSAIDs through a multiorifice catheter has the best effectiveness during the first 48 hours on postoperative pain intensity after elective cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* elective Cesarean Section under spinal anesthesia over37 weeks' gestation

Exclusion Criteria:

* allergy to NSAIDs
* ASA III or higher
* refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Cumulative intravenous morphine consumption | 48 hours

SECONDARY OUTCOMES:
Postoperative pain intensity at rest and mobilization | admission, 3,6,12,24,36,48h
adverse effects (nausea, vomiting, itching, sedation)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Cochin, Paris, France

REFERENCES:
- [Derived] Rackelboom T, Strat SL, Silvera S, Schmitz T, Bassot A, Goffinet F, Ozier Y, Beaussier M, Mignon A. Improving continuous wound infusion effectiveness for postoperative analgesia after cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2010 Oct;116(4):893-900. doi: 10.1097/AOG.0b013e3181f38ac6. PMID 20859153